CLINICAL TRIAL: NCT06814912
Title: Prospective Evaluation of Virtual Reality Headsets on Cancer Patients During Day Hospital Stay
Brief Title: Evaluation of Virtual Reality Headsets on Cancer Patients During Day Hospital Stay
Acronym: VIRTUEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Sainte Catherine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A01262-45
Record Dates: First submitted 2025-01-20; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- virtual reality headset (Experimental)
  Interventions: Other: Survey using a questionnaire

INTERVENTIONS:
Other: Survey using a questionnaire — virtual reality headset is added during treatment administration. Patient must complete a survey at the end of treatment administration and virtual headset use.

SUMMARY:
Use of virtula reality headsets during treatment course on day hospitalized cancer patients

ELIGIBILITY:
Inclusion Criteria:

* cancer patients
* chemotherapy treatment

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Rate of patients with nausea reduction compared with preview treatment administration | From the first chemotherapy injection until the end of chemotherapy injection with the virtual reality headset (at the end of the third cycle; each cycle is 21 days) )
  survey : improvement of nausea

CONTACTS AND LOCATIONS:
Locations (1):
- ICAP, Avignon, France

IPD SHARING:
Plan to Share IPD: No